CLINICAL TRIAL: NCT03830476
Title: Navigator ACT-Acceptance and Commitment Therapy-group Treatment for Distressed and Stressed Parents of Children with Disabilities
Brief Title: Navigator ACT Group Intervention for Parents of Children with Disabilities
Acronym: NavigatorACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Tatja Hirvikoski, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Navigator ACT
Record Dates: First submitted 2019-02-02; First posted 2019-02-05 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Parenting; Stress; Disability, Developmental; Behavior, Child; Acceptance and Action Processes; Parent-Child Relations; Experiential Avoidance; Depression, Anxiety
Keywords: Acceptance- and Commitment Therapy, ACT, parenting stress, parenting a child with disability, depression, anxiety, disabilities
MeSH Terms: conditions — Developmental Disabilities; Child Behavior; Depression; Anxiety Disorders | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Feasibility study and Randomised Controlled Trial
Who Masked: Care Provider
Masking Description: Masking at baseline of both participant and care-provider.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acceptance- and Commitment therapy group (Experimental): Experiment group that receives the treatment direct after the baseline measurement.
  Interventions: Behavioral: Acceptance- and Commitment therapy group for parents to children with disabilities
- Treatment as usual (Active Comparator): Comparison group that receives treatment as usual and the Navigator ACT intervention appr 6 months later.
  Interventions: Behavioral: Treatment as usual.

INTERVENTIONS:
Behavioral: Acceptance- and Commitment therapy group for parents to children with disabilities — ACT groups adjusted for parents of children with (any kind of) disabilities.
  Other Names: Navigator ACT group treatment
  Arms: Acceptance- and Commitment therapy group
Behavioral: Treatment as usual. — Treatment as usual within outpatient disability services.
  Arms: Treatment as usual

SUMMARY:
The main purpose of the pragmatic multicenter studies is to investigate the trransdiagnostic, manualized Acceptance and Commitment Therapy (ACT) based group treatment (Navigator ACT) for treatment of stress and distress in parents of children with disabilities, and to investigate the concept of parental psychological flexibility. The first phase includes a feasibility study (n=94) of the Navigator ACT for parents of children (0-17 years) with disabilties who participate in the Navigator ACT group treatment after being screened for symptoms of stress, depression and anxiety associated with the challenges of parenting. In the second phase (if treatment proves feasible), a randomised controlled trial (RCT) is conducted. In the RCT, approximately n=100 parents of children with disabilties were expected to be included, divided into experiment- and control groups. The recruitment takes places in several regions in Sweden. In addition, a psychometric evaluation of the main outcome instrument used in these studies, is going to be conducted. The Parental Acceptance and Action Questionnaire (PAAQ). In an additional study (expected n= ca 600), will focus on factors that explain treatment outcome and attrition.

DETAILED DESCRIPTION:
Navigator ACT group treatment is a novel, manual-based, transdiagnostic group treatment developed in Habilitation and Health, the disability services in the region Stockholm, in Sweden. The treatment consists of 5 sessions (each 3.5 hours), and has a main aim of increasing psychological flexibility of stressed and distressed parents raising a child with disability. The studies included in this project examine the feasibility and effectiveness of the manual-based Navigator ACT group treatment in the Swedish habilitation services context. The guestions we ask are; Is the Navigator ACT a feasible treatment in the disability services context? Is it effective in (a) improving parental psychological flexibility (b) increasing mindfulness (c) reducing symptoms of depression and anxiety (d) reducing parenting stress (e) reducing parent-reported difficulties ior increasing prosocial behaviors(e.g., behavioral problems) of children with disability.

FAS 1: The feasibility study is conducted in 7 disability service clinics in Stockholm and Uppsala, Sweden.The feasibility of Navigator ACT in the disability services context is measured by attendance, that is: parents participating in at least 4 out of 5 sessions are considered as completers. The parent and treatment provider satisfaction is measured by session- and course evaluations. Both parents and group leaders treatment credibility and expectancy is measured as well. Five self-rating questionnaires are used to measure efficacy: The Mindfulness Awareness Attention Scale (MAAS), Parental Acceptance and Action Questionnaire (PAAQ) Parental Stress Scale (PSS) Hospital Anxiety and depression scale (HADS), The Strengths and Difficulties Questionnaire (SDQ). Self-rating questionnaires are administered to parents at the baseline (0-2 weeks before the treatment start, T1), at the end of the treatment (0-2 weeks after, T2) and at the follow-up (3-4 months after the end of the treatment, T3). The data will be analyzed from baseline T1 to T2 (post treatment) as well as from T1 (baseline) to T3 (follow-up) with separate series of repeated measures ANOVA between-group.

FAS 2: Psychometric evaluation of the Parental Acceptance and Action Questionnaire (PAAQ).

FAS 2. The pragmatic multicenter RCT will be conducted in at least four regions of Sweden. Parents participating in the study have their children (0-17 years) currently enrolled in the disability services (experiment group n=42, control group n=42, totaling at least 84 parents, with the power calculation for medium large effect of 90% ES=0.50). To balance for attrition approximately 100 parents will be included in the study. The participants will be block randomized in several blocks. The experiment group will be receiving Navigator ACT treatment directly after the randomizing procedure, the Treatment-As-Usual (TAU) control group approximately six months after. The parents in the TAU group fill the effectiveness-related self-rating forms at the same measuring points as the parents in the experiment group as well during their own group process. The differences between the experiment and control groups will be analyzed by mixed-model linear regression.

FAS4: The aim of this study is reveal which parents get the most benefit of the Navigator ACT treatment, and what factors predict treatment competition vs. attrition.

The Regional Ethics Committee of Stockholm (2016/526-21-1,2016/115-31/4, 2017/573-31/5 ) has approved the studIes.

ELIGIBILITY:
Inclusion Criteria:

* a parent to a child 0-18 years with diagnosed disability
* mild to severe symptoms of parental stress, depression or anxiety
* a possibility to participate in all group sessions
* an ability to function in a group
* a knowledge of the Swedish language

Exclusion Criteria:

* deep depression with suicidality
* psychosis or manic episodes
* severe post-traumatic stress disorder (PTSD)
* homelessness or other extreme life situation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Parent report their own and their child's sex/gender during the screening interview.
Enrollment: 137 (Actual)
Dates: Start 2016-01-02 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
1. Change (increase) in parental psychological flexibility and experiential acceptance | [Time Frame: Change in psychological flexibility measured at baseline, immediately after the intervention and at three-four month follow-up]
  Parental Acceptance and Action Questionnaire (PAAQ), a scale that targets psychological flexibility and experiential acceptance in the parenting context, i.e. measures to which extent parents' accept inner experiences related to parenting and the readiness to take appropriate/needed action in parenting (commitment to values-based actions). Originally 19-item scale.

SECONDARY OUTCOMES:
2. Change (increase) in mindfulness skills | [Time Frame: Change in psychological flexibility measured at baseline, immediately after the intervention and at three-four month follow-up]
  The Mindfulness Awareness Attention Scale (MAAS), a 15-item scale (scored 1-6) assessing dispositional mindfulness in regards to cognitive, emotional, physical, interpersonal and general domains.
3. Change (decrease) in depression and anxiety | [Time Frame: Change in psychological flexibility measured at baseline, immediately after the intervention and at three-four month follow-up]
  Hospital Anxiety and Depression Scale (HADS). Has 14 items scored 0 ("Often") - 3 ("Seldom"), subsequently summarized for an overall score; high scores indicate higher levels of depression or anxiety.
4. Change (decrease) in parental stress. | [Time Frame: Change in psychological flexibility measured at baseline, immediately after the intervention and at three-four month follow-up]
  The Parental Stress Scale (PSS) is a18-item tool for measurement of parenting stress, scored 1-5 on a 5-point Likert scale. The initial factor has suggested four-factor structure for the PSS consisting of parental 1) rewards, 2) stressors, 3) lack of control and 4) satisfaction in parenting. High scores indicate higher levels of stress in parenting context.
5. Change (decrease) in child's difficulties and the impact of these difficulties on the child's family. | [Time Frame: Change in psychological flexibility measured at baseline, immediately after the intervention and at three-four month follow-up]
  The Strengths and Difficulties Questionnaire (P4-17 SDQ), a caregiver administered, 25-item extended version of SDQ used for behavior screening of children and adolescents in ages 4-17 years. The SDQ P4-17 covers common areas of emotional and behavioral difficulties and strengths as well as includes a caregiver reported impact- and burden assessment.

OTHER OUTCOMES:
Treatment Credibility Scale (TCS) | Measured at baseline,and immediately after the intervention.
  As a measure of feasibility, TCS is used to measure the expectation of improvement and treatment credibility. The TCS is a visual analogue scale rated from "Low credibility"/ "Not at all" (0) to "High credibility"/"Very much" (10) and the score calculated is a mean of all items. The TCS was administered after providing thorough information and presentation of the treatment content at baseline and after completion of the treatment. The item wording after adjustment to the current study were: (1) How logical does Navigator ACT treatment seem to you? (2) How confident are you that this treatment will reduce your distress? (3) Would you recommend Navigator ACT to a friend experiencing the same type of distress? (4) How successful do you feel this type of intervention is in improving your psychological health? 5) At this very moment, to what degree the intervention has improved your psychological health?
Session Evaluation Form (SEF) | Up to 3 months
  Measures treatment satisfaction regarding each treatment session
Patient Evaluation Form (PEF) | Up to 3 months
  Measures overall treatment satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- Tiina Maria Holmberg Bergman, Knivsta, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Acceptance and Commitment Therapy Group Intervention for Parents of Children with Disabilities (Navigator ACT): An Open Feasibility Trial — https://link.springer.com/content/pdf/10.1007/s10803-022-05490-6.pdf